CLINICAL TRIAL: NCT01281579
Title: An Open-Label, Randomized, Parallel-Group, Single-Center Study to Evaluate the Single and Multiple Dose Pharmacokinetic and Pharmacodynamic Characteristics of JNJ-28431754 (Canagliflozin) in Healthy Subjects
Brief Title: A Single and Multiple Dose Study of Canagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017695; 28431754DIA1030
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics; Canagliflozin
MeSH Terms: interventions — Canagliflozin

ARMS (3):
- 001 (Experimental): Canagliflozin 50 mg Tablets oral 50-mg once daily on Day 1 and on Days 4 through 9.
  Interventions: Drug: Canagliflozin 50 mg
- 002 (Experimental): Canagliflozin 100 mg Tablets oral 100-mg once daily on Day 1 and on Days 4 through 9.
  Interventions: Drug: Canagliflozin 100 mg
- 003 (Experimental): Canagliflozin 300 mg Tablets oral 300-mg once daily on Day 1 and on Days 4 through 9.
  Interventions: Drug: Canagliflozin 300 mg

INTERVENTIONS:
Drug: Canagliflozin 100 mg — Tablets, oral, 100-mg, once daily on Day 1 and on Days 4 through 9.
  Arms: 002
Drug: Canagliflozin 50 mg — Tablets, oral, 50-mg, once daily on Day 1 and on Days 4 through 9.
  Arms: 001
Drug: Canagliflozin 300 mg — Tablets, oral, 300-mg, once daily on Day 1 and on Days 4 through 9.
  Arms: 003

SUMMARY:
The purpose of this study is to determine blood and urine concentrations of canagliflozin and glucose in healthy adult volunteers after administration of single and multiple doses of canagliflozin.

DETAILED DESCRIPTION:
This is an open-label (volunteers and study staff will know the name and dose of the treatment assigned), single-center study of canagliflozin (JNJ-28431754) in healthy adult volunteers. Canagliflozin (a sodium-glucose cotransporter 2-inhibitor) is currently under development to lower blood sugar levels in patients with Type 2 diabetes mellitus (T2DM). Healthy volunteers will take canagliflozin 50 mg, 100 mg, or 300 mg tablets, orally (by mouth), once daily on Day 1 and on Days 4 to 9. All study drug administration will occur at approximately the same time each morning with 240 mL of noncarbonated water and will be followed by a standardized breakfast within 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 18 and 30 kg/m2, inclusive, and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to drugs or lactose
* Known allergy to canagliflozin or any of the excipients of the formulation of canagliflozin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | At protocol-specified times up to Day 14
Urine concentrations of canagliflozin | At protocol-specified times up to Day 11
Plasma glucose concentrations | At protocol-specified times up to Day 11
Urine glucose concentrations | At protocol-specified times up to Day 11

SECONDARY OUTCOMES:
The number and type of adverse events reported | Up to 10 days after last dose" (last dose is given on Day 9)
Changes in hematology, chemistry and urinalysis parameters | Up to 10 days after last dose" (last dose is given on Day 9)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.